CLINICAL TRIAL: NCT06987617
Title: Pilot Study to Investigate the Impact of an App on the Quality of Life and Symptoms of Individuals Affected by Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endo Health GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RCT_PilotMeno
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Menopausal and Other Perimenopausal Disorders
Keywords: Menopause; Digital Therapeutics; Quality of Life

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group has access to the menopause app and its functions in addition to care-as-usual
  Interventions: Device: Menopause App
- Control Group (No Intervention): Control group has access to care-as-usual only

INTERVENTIONS:
Device: Menopause App — The menopause app facilitates the implementation of multimodal self-management strategies in the daily routines of individuals with a (peri-)menopausal disorder, through tools such as a symptom diary and guided interactive exercises.
  Arms: Intervention Group

SUMMARY:
The study explores the impact of a digital app for the self-management of (peri-)menopausal disorders. A total of 224 participants were randomized into an intervention and a control group. Findings indicate that the app offers beneficial effects on menopausal symptoms and menopause-specific quality-of-life. The study also provided valuable insights for the design of future larger trials and highlights the promising potential of the app to enhance individualized care.

ELIGIBILITY:
Inclusion Criteria:

* Legal capacity
* Residency in Germany
* Female sex
* Age ≥18 years
* Known and medically confirmed (peri-)menopausal disorder (N95.1, N95.3, N95.8, N95.9)
* Ownership of a smartphone and ability to use it
* Internet access for app usage and questionnaire completion
* Email address for registration
* Willingness to complete questionnaires online
* Motivation for regular app usage
* Sufficient proficiency in the German language
* Absence of exclusion criteria

Exclusion Criteria:

* Changes in hormone therapy within eight weeks before the start of the study and/or planned within the next 12 weeks
* Changes in antidepressant treatment within eight weeks before the start of the study and/or planned within the next 12 weeks
* Previous or current access to the Endo-App or other comparable digital health applications, or current active prescription
* Current participation in other clinical studies
* Failure to meet the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Menopause-specific Quality of Life Questionnaire (MENQOL) | From enrollment (baseline) to the end of treatment at 12 weeks
  Menopause-specific Quality of Life Questionnaire (MENQOL): Min=1, max=8. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Endo Health GmbH, Chemnitz, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No